CLINICAL TRIAL: NCT05719194
Title: Effect of a Personalized Weaning Strategy on Weaning Success
Acronym: P-Wean
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: P-Wean PHRC IR 2020 AUDARD
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Weaning; Mechanical Ventilation; Intubation
Keywords: WIPO; Extubation; Spontaneous Breathing Trial; T-piece; Pressure Support Ventilation; Weaning strategy; Personalization
MeSH Terms: interventions — Serum Bactericidal Test

STUDY DESIGN:
Intervention Model Description: Pragmatic, controlled, multicenter, stepped wedge cluster randomized trial, considering centers as clusters.
Who Masked: Outcomes Assessor
Masking Description: Double blind is not possible as this study evaluate a care strategy. However, in order to limit evaluation bias, the methodologist will be blinded to the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard intervention (Active Comparator)
  Interventions: Other: Standard SBT
- Personalized intervention - WIPO risk factors vs no risk factors (Experimental)
  Interventions: Other: SBT with T-piece or PSV

INTERVENTIONS:
Other: Standard SBT — Weaning strategy in accordance with the care practices of the department, regarding the assessment of weaning criteria, SBT and extubation modalities.
  Arms: Standard intervention
Other: SBT with T-piece or PSV — - Risk factors of WIPO
  Step 1 : Daily assessment of weaning criteria in accordance with the study protocol.
  Step 2 : Spontaneous breathing trial with T-piece for an hour. Measure of protein and haemoglobin by blood sample before and after the trial.
  Step 3 : Reconnect the patient to the ventilator for at least 30 minutes and then extubate if SBT is successful.
  If SBT failed : no extubation and new SBT the next day. Optimization of cardiac function or fluid overload will be in charge of the investigator.
  - No risk factors of WIPO
  Step 1 : Daily assessment of weaning criteria in accordance with the study protocol.
  Step 2 : Spontaneous breathing trial with pressure support ventilation (pressure support from 5 to 8 cmH20 - PEEP at 0 cmH20) for an hour.
  Step 3 : Reconnect the patient to the ventilator for at least 30 minutes and then extubate if SBT is successful.
  Arms: Personalized intervention - WIPO risk factors vs no risk factors

SUMMARY:
Weaning from mechanical ventilation is a daily challenge in intensive care units, as it can take up to 50% of the total duration of ventilation. The longer the duration of ventilation is, the more there is complication related with it.

Even when the spontaneous breathing trial is succeeded, 10 to 20% of extubations are failed and requires re-intubation.

There is two different ways to assess if the patient is capable of breathing by its own : T-piece which can be considered as hard to succeed (it can delay extubation for some patients) or pressure support ventilation with no PEEP which can be too easy and lead to an extubation too early.

Studies have identified risk factors of weaning induced pulmonary oedema wich is one of the main cause of failed extubation (up to 60%).

The purpose of P-WEAN is to evaluate whether a personalized strategy for weaning from mechanical ventilation, including daily search for weaning criteria and individualization of the weaning modality (T-piece or pressure support ventilation with zero PEEP) based on the existence of WIPO risk factors (obesity, COPD, heart disease) improves weaning success compared with usual practice.

DETAILED DESCRIPTION:
Before the study begin, all participating centers will be randomized to determine the time between the control and the interventional period. Patients included in the study will not be randomized individually but will be managed either according to the standard of care of the service or according to the personalized strategy (according to the stepped wedge group of the center).

* Control period: Patients will be subjected to a weaning strategy in accordance with the usual care practices of the service (evaluation of the criteria of weanability, the modalities of the spontaneous breathing trial and extubation)
* Interventional period: Patients will undergo a protocolized and standardized weaning strategy, including a daily assessment of weaning criteria, and a weaning trial (PSV or T-piece) whose modalities will be defined by the presence or the absence of weaning induced pulmonary oedema risk factors. These are :
* Obesity defined as BMI greater than 30 kg/m²
* Suspected or known COPD
* Heart disease whether it is structural (hypertrophic, dilated, valvular), functional (diastolic or systolic dysfunction), ischemic, or dysrhythmic.

Step 1 :

Daily assessment of weaning criteria in accordance with the study protocol

Step 2 :

* No risk factors : spontaneous breathing trial for 1 hour with pressure support ventilation (setting a pressure support level of 5 to 8 cm of water with no PEEP)
* Risk factors : spontaneous breathing trial with a T-piece for 1 hour, measuring protein and hemoglobin by blood sample before and after the trial.

Step 3 : Reconnecting the patient for at least 30 minutes and extubation if the SBT is successful. If not, the optimization of cardiac function or fluid overload will be the responsibility of the clinician.

Decisions regarding the use of non-invasive ventilation (NIV) or high-flow nasal oxygenation, will be made based on each centre's expertise and current clinical practice to minimize interference with the study procedure. However, knowing the recent data and the possible superiority of NIV in preventing post-extubation respiratory failure for high risk patients, investigators will be strongly encouraged to prioritize the prophylactic use of NIV (over high-flow nasal oxygenation) after tracheal extubation.

Patients will be assessed by members of the investigating center's research team (under the supervision of the centre's investigators) at least daily during hospitalization in the ICU and until day 28 post-randomization, as well as at discharge and at 90 days.

ELIGIBILITY:
Inclusion Criteria : all patients ≥ 18 y.o admitted to the ICU, under invasive mechanical ventilation for more then 24 hours and fullfilling the following weaning criteria :

* Resolution or improvement of the condition that led to intubation, as judged by the clinician in charge of the patient.
* Hemodynamic stability, defined as systolic blood pressure between 90 and 160 mmHg, heart rate less than 140 beats/min, without or with low doses of vasopressors.
* Glasgow score of 13 or greater and Richmond Agitation-Sedation Scale (RASS) score between -1 and +1.
* Respiratory stability defined as: oxygen saturation > 90% with inspired oxygen fraction ≤ 0.5 and PEEP ≤ 8 cmH2O, respiratory rate < 35/min, spontaneous tidal volume > 5 mL/kg, and peak inspiratory pressure ≤ 15 cmH2O.
* Few secretions (< 3 aspirations in the past 8 hours).
* Effective cough.
* Negative leak test (>100 mL or >10%).
* No surgery planned within 72 hours.
* Patients with a social security plan.

Exclusion Criteria:

* Acute cerebral pathology requiring admission to intensive care and/or mechanical ventilation with tracheal intubation for neurological reasons (Glasgow score <13 at the time of intubation or CT scan abnormality): hemorrhagic stroke without or with vascular malformation (aneurysm, arterio-venous malformation...), ischemic stroke, head trauma, cerebral anoxo-ischemia after cardiac arrest.
* Tetraplegic or paraplegic patients with lesion level higher than D8.
* Peripheral neuromuscular pathology (underlying myopathy or myasthenia).
* ICU's Neuromyopathy.
* Tracheostomy.
* Patients with a decision of non-reintubation or terminal intubation.
* Pregnant or lactating women.
* Patients already included in this study.
* Patients under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Mortality at day 28, reintubation at 72 hours, ventilatory free days (VFDs) from first spontaneous breathing trial to day 28. | 28 days
  Composite score including those three criteria such that mortality is a more severe outcome than reintubation and the number of VFDs, and reintubation is a more severe outcome than the number of VFDs

SECONDARY OUTCOMES:
Rate of extubation success after the first SBT. | 72 hours from first SBT
Rate of reintubation | 72 hours from first SBT
Rate of reintubation | 72 hours from extubation
Reintubation rate within 7 days of extubation. | 7 days after extubation
Time from first SBT to extubation. | 28 days
SBT failure rate | 28 days
  Defined by respiratory rate increase of 50% or > 35/min, dyspnea, SpO2 < 88% or decrease of 5%, heart rate increase > 20%, systolic blood pressure increase > 20%, agitation, sweating.
Number of days without mechanical ventilation | From day one of first SBT to day 28
Length of stay in the ICU and in the hospital. | 90 days
Mortality of ICU stay/hospital stay. | 90 days
Mortality at day 28. | 28 days
Mortality at day 90. | 90 days

OTHER OUTCOMES:
Rate of tracheostomy during the ICU stay. | 28 days
Incidence of non-invasive ventilation or high-flow nasal oxygenation post-extubation, both prophylactic and curative. | 72 hours after extubation.
Incidence of use for diuretics or beta-blockers for failed weaning trials or WIPO. | 28 days
Incidence of the absence of extubation despite a successful SBT. | 28 days
Time and reason for reintubation in case of failed extubation. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jules Audard, Study Chair — CHU de Clermont-Ferrand
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Lyon - Hôpital Lyon Sud, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse